CLINICAL TRIAL: NCT01639300
Title: Randomised Placebo-Controlled Single Blind Study to Investigate Single Ascending Doses of GNbAC1 in Multiple Sclerosis Patients Followed by Open-label Extension With Repeated Doses of GNbAC1
Brief Title: Safety Study of GNbAC1 in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GeNeuro Innovation SAS (Industry)
Responsible Party: Sponsor
Organization: GeNeuro SA (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GNC-002
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Forms of Multiple Sclerosis; Progressive Forms of Multiple Sclerosis; GNbAC1; Monoclonal antibody; Multiple Sclerosis Associated Retrovirus (MSRV); Temelimab
MeSH Terms: conditions — Multiple Sclerosis | interventions — temelimab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GNbAC1 (Experimental)
  Interventions: Biological: GNbAC1
- GNbAC1 placebo (Placebo Comparator)
  Interventions: Biological: GNbAC1 placebo

INTERVENTIONS:
Biological: GNbAC1 — Single dose intravenous (IV) GNbAC1 2mg/kg or 6mg/kg
  Arms: GNbAC1
Biological: GNbAC1 placebo — Single dose intravenous (IV) GNbAC1 placebo
  Arms: GNbAC1 placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of single ascending doses, as well as of repeated administrations of GNbAC1 in MS patients.

Scientific research has shown that the expression of genes of a virus which is integrated in the Human genetic material, the Multiple Sclerosis associated RetroVirus (MSRV) could play a critical role in the causation of multiple sclerosis.

GNbAC1 is an experimental medication, which neutralizes (i.e. inactivates) a protein of MSRV that might contribute to the development or deterioration of multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients (if female, neither pregnant nor breast-feeding, should be post-menopausal or surgically sterile, or should use two highly effective method of contraception such as oral contraception plus mechanical barrier); Male subjects with partners of childbearing potential have to use adequate contraception during the study. Contraception methods should be followed during the study and up to 3 months after the last study drug administration. Female subjects who are women of childbearing potential (WOCBP) will have to be tested negative with a pregnancy test (serum or urine) at screening and Day 1 and before each repeated administrations of GNbAC1.
* Between 18 and 65 years of age;
* Patients with Primary Progressive MS (PPMS) according to the Revised McDonald criteria 2010 or patients with Secondary Progressive MS (SPMS) or patients with Relapsing-Remitting MS(RRMS)according to the Revised McDonald criteria 2010 who cannot be treated with available treatments for MS due to intolerance, non response or refusal of treatment;
* Score ≤ 6.5 on the Expanded Disability Status Scale (EDSS);
* Body weight between 40 and 100kg.

Exclusion Criteria:

* Positive serology for viral hepatitis and HIV;
* Disease other than MS that could better explain his/her signs and symptoms;
* Previously treated with cladribine, lymphoid irradiation or depleting antibodies;
* Usage in the last 3 months of interferon beta or glatiramer acetate;
* Any usage in the last 6 months of mitoxantrone, cytotoxic immunosuppressive therapy, natalizumab, fingolimod or immunoglobulin;
* Usage within 30 days prior to baseline of oral or systemic corticosteroids or ACTH;
* Inadequate liver function;
* Severe renal impairment;
* Severe psychiatric disorder;
* Known inability to undergo an MRI scan;
* Having participated in another clinical study within 6 months prior to study baseline except for patients who have participated or who are currently participating in an interventional study without any study drug intake.
* Pregnancy or breastfeeding
* Female subjects considering becoming pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of single ascending doses, as well as of repeated administrations of GNbAC1 in MS patients. | 177 days

SECONDARY OUTCOMES:
To determine the pharmacokinetics (PK) characteristics following administration of single ascending doses, as well as of repeated administrations, of GNbAC1 in MS patients | 177 days
To determine pharmacodynamic markers of MS disease activity in patients including measurement of MSRV-Env markers and magnetic resonance imaging (MRI) | 177 days
To assess the immunogenicity of GNbAC1. | 177 days

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Derfuss, MD, Principal Investigator — University Hospital, Basel, Switzerland; Patrice Lalive, MD, Principal Investigator — HUG
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel
  - Hopitaux Universitaires de Genève - HUG, Geneva

REFERENCES:
- [Derived] Derfuss T, Curtin F, Guebelin C, Bridel C, Rasenack M, Matthey A, Du Pasquier R, Schluep M, Desmeules J, Lang AB, Perron H, Faucard R, Porchet H, Hartung HP, Kappos L, Lalive PH. A phase IIa randomised clinical study of GNbAC1, a humanised monoclonal antibody against the envelope protein of multiple sclerosis-associated endogenous retrovirus in multiple sclerosis patients. Mult Scler. 2015 Jun;21(7):885-93. doi: 10.1177/1352458514554052. Epub 2014 Nov 12. PMID 25392325
- See also: MedlinePlus related topics: Multiple Sclerosis — http://www.nlm.nih.gov/medlineplus/multiplesclerosis.html
- See also: MedlinePlus related topics: Multiple Sclerosis — https://www.ncbi.nlm.nih.gov/pubmed/26198921